CLINICAL TRIAL: NCT06147297
Title: Using Music to Promote Young People's Emotion Regulation and Reduce Their Depressive and Anxious Symptoms and Loneliness: A Pilot Randomised Controlled Trial
Brief Title: Music Program for Hong Kong Adolescents: Improving Emotion Regulation and Reducing Depression, Anxiety, and Loneliness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Queensland (Other); The Hong Kong Polytechnic University (Other); Health and Medical Research Fund (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EA230395; 10211636 (Other Grant/Funding Number: Health and Medical Research Fund)
Record Dates: First submitted 2023-11-19; First posted 2023-11-27 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Emotion Regulation; Depressive Symptoms; Anxiety; Loneliness
Keywords: Adolescence; Youth; Emotion Regulation; Music; Loneliness; Mental Health; Psychoeducation
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Intervention group: Receive the music-based program, and complete the survey before- and after- the program.
  Waitlist group: Invited to complete the survey before- and after the 4-week waiting period. Then the waitlist group will also be offered the program, and invited to complete an optional post-program survey.
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Receive the music-based program once a week for 4 weeks, each session is 60 to 90 minutes, and participants will complete the survey before- and after- the program.
  Interventions: Behavioral: Tuned In
- Wait-list group (No Intervention): Complete the survey before- and after the 4-week waiting period. Then the waitlist group will also be offered the program, and invited to complete an optional post-program survey

INTERVENTIONS:
Behavioral: Tuned In — The Tuned In programme is based on Russell's (1980) circumplex model of emotion, which categories emotions along the two dimensions of valence and arousal. Through psychoeducation and group discussions, participants in the programme first learn how to categorise their emotions in terms of intensity (i.e., arousal level) and positivity (i.e., valence). They then reflect on and develop a list of songs that they relate to personally and use them to increase or decrease the intensity and positivity of their emotions. In other words, the participants practise monitoring their emotional state and use music to help them modify how they feel. The programme will be conducted by a facilitator with a psychology background, and a registered music therapist.
  Arms: Intervention group

SUMMARY:
This study is a clinical trial that aims to test and validate a music-based program called "Tuned In" in helping adolescents in Hong Kong improve their mental well-being. The researchers want to find out if the program can help participants enhance their ability to regulate their emotions, reduce mood symptoms and feelings of loneliness.

Participants in the study will be randomly assigned to either the group that receives the program right away (intervention group) or the group that waits for four weeks before receiving the program (wait list group). They will take part in a group-based weekly program for four weeks. Additionally, they will be asked to complete questionnaires before and after the program to see if there are any changes in their mental well-being. The program will be delivered by a facilitator with a psychology background, and a registered music therapist.

By addressing the gaps in mental health interventions for young people in Hong Kong, this study aims to contribute to the development of effective strategies to support their emotional well-being.

ELIGIBILITY:
Inclusion Criteria:

* self-report as having problems with low mood, anxiety or loneliness
* score 3 or above on the General Health Questionnaire (GHQ-12), which indicates psychological distress.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-08-17 (Estimated); Study Completion 2025-08-17 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Skills | Questionnaires will be administered before the start of the program, and immediately after the program (intervention group) or after 4 weeks of wait period (wait-list group)
  To assess difficulties, strategies, and confidence in emotion regulation, we will use the Emotion Regulation Questionnaire (Liu et al., 2015), Difficulties in Emotion Regulation scale, and select items from Dingle and Carter's (2017) program evaluation tool.

SECONDARY OUTCOMES:
Mood symptoms | Questionnaires will be administered before the start of the program, and immediately after the program (intervention group) or after 4 weeks of wait period (wait-list group)
  The Depression Anxiety Stress Scale-21 (Moussa et al., 2001; DASS-21) will be used to measure mood symptoms
Loneliness | Questionnaires will be administered before the start of the program, and immediately after the program (intervention group) or after 4 weeks of wait period (wait-list group)
  The Hong Kong version of the De Jong Gierveld Loneliness Scale (Leung et al., 2008) will be used to measure loneliness

OTHER OUTCOMES:
Anhedonia | Questionnaires will be administered before the start of the program, and immediately after the program (intervention group) or after 4 weeks of wait period (wait-list group)
  The Chinese version of the Snaith-Hamilton-Pleasure scale (Liu et al., 2012) will be used to measure anhedonia.
Program acceptability and feasibility | Questionnaire will be administered immediately after the program
  Furthermore, we plan to examine the acceptability of the program with the Hong Kong adolescents. This will be done using a combination of quantitative and qualitative approaches. Satisfaction ratings will be collected from the participants, on a 7-point Likert scale. The questions will be on the perceived usefulness of the program, the level of interest in the program, the likelihood of them recommending the program to other adolescents, and the likelihood of them to continue using music as an emotion regulatory strategy in the future (Dingle et al., 2016). We will also use open-ended questions to obtain feedback from the participants on their experiences of the program, and ask for suggestions for improvements for a future RCT. Furthermore, as feasibility indicators, we will also record the recruitment rate and dropout rate of this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Cao, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Dingle GA, Carter NA. Smoke into Sound: A pilot randomised controlled trial of a music cravings management program for chronic smokers attempting to quit. Musicae Scientiae. 2017 Jun;21(2):151-77.
- [Background] Dingle GA, Fay C. Tuned In: The effectiveness for young adults of a group emotion regulation program using music listening. Psychology of Music. 2017 Jul;45(4):513-29.
- [Background] Dingle GA, Hodges J, Kunde A. Tuned In Emotion Regulation Program Using Music Listening: Effectiveness for Adolescents in Educational Settings. Front Psychol. 2016 Jun 7;7:859. doi: 10.3389/fpsyg.2016.00859. eCollection 2016. PMID 27375537
- [Background] Dingle GA, Sharman LS, Bauer Z, Beckman E, Broughton M, Bunzli E, Davidson R, Draper G, Fairley S, Farrell C, Flynn LM, Gomersall S, Hong M, Larwood J, Lee C, Lee J, Nitschinsk L, Peluso N, Reedman SE, Vidas D, Walter ZC, Wright ORL. How Do Music Activities Affect Health and Well-Being? A Scoping Review of Studies Examining Psychosocial Mechanisms. Front Psychol. 2021 Sep 8;12:713818. doi: 10.3389/fpsyg.2021.713818. eCollection 2021. PMID 34566791
- [Background] Hutchison AN, Yeung DY, Gerstein LH, Wettersten KB. Psychometric comparison of Chinese and English versions of the Emotion Regulation Questionnaire with bilingual Hong Kong Chinese students. Int J Psychol. 2021 Apr;56(2):296-303. doi: 10.1002/ijop.12699. Epub 2020 Jul 23. PMID 32700781
- [Background] Leung GT, de Jong Gierveld J, Lam LC. Validation of the Chinese translation of the 6-item De Jong Gierveld Loneliness Scale in elderly Chinese. Int Psychogeriatr. 2008 Dec;20(6):1262-72. doi: 10.1017/S1041610208007552. Epub 2008 Jul 1. PMID 18590603
- [Background] Leung MC, Cheung RY. Music engagement and well-being in Chinese adolescents: Emotional awareness, positive emotions, and negative emotions as mediating processes. Psychology of Music. 2018;48(1):105-19.
- [Background] Li J, Han ZR, Gao MM, Sun X, Ahemaitijiang N. Psychometric properties of the Chinese version of the Difficulties in Emotion Regulation Scale (DERS): Factor structure, reliability, and validity. Psychol Assess. 2018 May;30(5):e1-e9. doi: 10.1037/pas0000582. PMID 29756796
- [Background] Li X, Shek DTL, Shek EYW. Psychological Morbidity among University Students in Hong Kong (2014-2018): Psychometric Properties of the Depression Anxiety Stress Scales (DASS) and Related Correlates. Int J Environ Res Public Health. 2021 Aug 5;18(16):8305. doi: 10.3390/ijerph18168305. PMID 34444053
- [Background] Liu W, Chen L, Tu X. Chinese adaptation of Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CCA): A psychometric evaluation in Chinese children. Int J Psychol. 2017 Oct;52(5):398-405. doi: 10.1002/ijop.12233. Epub 2015 Nov 26. PMID 26611865
- [Background] Liu WH, Wang LZ, Zhu YH, Li MH, Chan RC. Clinical utility of the Snaith-Hamilton-Pleasure scale in the Chinese settings. BMC Psychiatry. 2012 Oct 31;12:184. doi: 10.1186/1471-244X-12-184. PMID 23110667
- [Background] Moussa MT, Lovibond PF, Laube R. Psychometric properties of a Chinese version of the short Depression Anxiety Stress Scales (DASS21). Report for New South Wales Transcultural Mental Health Centre, Cumberland Hospital, Sydney. 2001.
- [Background] Remmington NA, Fabrigar LR, Visser PS. Reexamining the circumplex model of affect. J Pers Soc Psychol. 2000 Aug;79(2):286-300. doi: 10.1037//0022-3514.79.2.286. PMID 10948981
- [Derived] Cao Y, Shi Y, Low DCW, Shek DTL, Shum DHK, Tanksale R, Dingle G. Using Music to Promote Hong Kong Young People's Emotion Regulation and Reduce Their Mood Symptoms and Loneliness: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 16;14:e67764. doi: 10.2196/67764. PMID 40239199